CLINICAL TRIAL: NCT05686915
Title: Metal Artifact Reduction Sequence MRI in Revision Total Hip Arthroplasty With a Ceramic Femoral Head and Titanium Sleeve
Brief Title: MARS MRI in Revision THA With a Ceramic Femoral Head and Titanium Sleeve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Jason Jennings, Orthopedic Surgeon, Colorado Joint Replacement
Other Study IDs: 1969400
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Revision; Titanium Sleeve

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Revision Total Hip Arthroplasty: Patients who received a revision total hip surgery utilizing a ceramic femoral head with a titanium sleeve
  Interventions: Diagnostic Test: MARS MRI; Diagnostic Test: Titanium Labs; Diagnostic Test: Cobalt Labs; Diagnostic Test: Chromium Labs

INTERVENTIONS:
Diagnostic Test: MARS MRI — metal artifact reduction sequence (MARS) MRI to assess for fluid collections, ATLRs or other abnormalities
Diagnostic Test: Titanium Labs — Labs to look at titanium levels in blood
Diagnostic Test: Cobalt Labs — Labs to look at cobalt levels in blood
Diagnostic Test: Chromium Labs — Labs to look at chromium levels in blood

SUMMARY:
Revision total hip replacement using a ceramic head utilizes a titanium sleeve which introduced another articulation into the system that may lead to a local soft tissue reaction. The purpose of this study is to determine the frequency, size and types of MRI documented local tissue reactions in individuals doing well after a revision total hip replacement and ceramic bearing surface that utilizes a titanium sleeve.

DETAILED DESCRIPTION:
Metal-on-metal total hip arthroplasty (THA) were heralded as a solution for two of the most common problems in hip arthroplasty in the last decade, instability and osteolysis. Unfortunately, their failures have led to diminished enthusiasm for this bearing surface. Adverse local tissue reactions (ATLRs) have been well documented as a means of pain and failure in this population. A recent report revealed that the most commonly used bearing surface in total hip arthroplasty, metal-on-polyethylene, may have up to a 28% incidence of MRI abnormalities in asymptomatic hips. Revision THA using a ceramic head utilizes a titanium sleeve which introduced another articulation into the system that may lead to a local soft tissue reaction. The purpose of this study is to determine the frequency, size and types of MRI documented local tissue reactions in asymptomatic individuals after a revision THA and ceramic bearing surface that utilizes a titanium sleeve. To our knowledge, this has not been studied previously and may provide important baseline features of this diagnostic tool with this particular bearing surface. We hypothesize that there will be fluid collections in a small but clinically significant portion of asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a revision total hip surgery utilizing a ceramic femoral head with a titanium sleeve
* Patient whose age ranges from 18-99
* Patients who are not experiencing groin pain, thigh pain, or pain with ROM of the hip
* Patients who are at least 2 years after a revision THA
* Acetabular implant (cup) was placed in the appropriate position
* Patients with a Harris Hip Score of >90

Exclusion Criteria:

* Patients who do not meet the above criteria
* Patients unable to have an MRI (i.e. pacemaker, metal implants or issues with claustrophobia requiring sedation)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a revision total hip surgery utilizing a ceramic femoral head with a titanium sleeve
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
MARS MRI abnormalities | 2 Years Post Revision Total Hip Replacement
  Local Tissue Reactions or Fluid collections on the MARS MRI Scan

SECONDARY OUTCOMES:
Titanium Lab Value | 2 Years Post Revision Total Hip Replacement
  Titanium levels in blood
Chromium Lab Value | 2 Years Post Revision Total Hip Replacement
  Chromium levels in blood
Cobalt Lab Value | 2 Years Post Revision Total Hip Replacement
  Cobalt levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Jennings, MD, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fehring TK, Fehring K, Odum SM. Metal artifact reduction sequence MRI abnormalities occur in metal-on-polyethylene hips. Clin Orthop Relat Res. 2015 Feb;473(2):574-80. doi: 10.1007/s11999-014-3873-6. PMID 25141843